CLINICAL TRIAL: NCT02985502
Title: The Comparison and Association of Fatigue, Self-care Activities and Quality of Life in Patients With Pancreatogenic Diabetes Mellitus After Total Pancreatectomy or Pancreaticoduodenectomy
Brief Title: The Comparison of Quality of Life in Patients With Pancreatogenic Diabetes After Pancreatectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201611038RINB
Record Dates: First submitted 2016-12-05; First posted 2016-12-07 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Quality of Life; Diabetes Mellitus; Pancreatectomy
Keywords: Quality of Life; Diabetes Mellitus; Pancreatectomy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- pancreatogenic diabetes: patients with pancreatogenic diabetes after pancreatectomy will be recruited
  Interventions: Other: pancreatogenic diabetes

INTERVENTIONS:
Other: pancreatogenic diabetes — pancreatogenic diabetes

SUMMARY:
Background: Pancreatogenic diabetes resulted from total pancreatectomy(TP) is one of the reason why this form of surgery technique is seldom performed. However, with the progress of medical and surgical care nowadays, patients undergone TP could receive better care in endocrine and exocrine insufficiency. In addition, with better understanding of benign pancreatic tumors and pancreatic neuroendocrine tumors, more patients with diffused pancreatic disease are diagnosed; hence, the performance of TP may rise. Nevertheless, the quality of life of patients with pancreatogenic diabetes after TP is still currently controversial.

Purpose: The purpose of this study is to (1) explore the association of fatigue, self-care activities and quality of life in patients with pancreatogenic diabetes after total pancreatectomy; (2) compare the data with diabetic patients after pancreaticoduodenectomy.

Method: A correlational and comparative cross-sectional approach will be used. The data will be collected with a structured questionnaire via purposive sampling of 120 subjects in an outpatient pancreatic surgical department. Inclusion criteria will be the patients with: (1) age 20 or above, (2) conscious clear, can communicate in Mandarin or Taiwanese, (3) agree to participate in the study and sign informed consent. Exclusion criteria will be the patients diagnosed with cancer other than pancreatic cancer and under active treatment. Data will go through propensity score matching and will be analyzed by using descriptive statistics, paired t-test, Chi square test, Pearson's correlation, and conditional logistic regression.

Anticipated achievement: The anticipated achievement of this study is to understand the relationships between fatigue, self-care activities, and quality of life in patients with pancreatogenic diabetes after pancreas surgery. In addition, through this study, the influence of diabetes to patients after pancreatic tumor resection can be explored; and the factors that influence the population's quality of life can be examined. By the filling of this knowledge gap, intervention can be planned accordingly to help improve the population's quality of life.

ELIGIBILITY:
Inclusion Criteria:

* (1) age 20 or above, (2) conscious clear, can communicate in Mandarin or Taiwanese, (3) agree to participate in the study and sign informed consent

Exclusion Criteria:

* diagnosed with cancer other than pancreatic cancer and under active treatment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with pancreatogenic diabetes after total pancreatectomy or pancreaticoduodenectomy
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Questionnaire | 1 day at first appointment

CONTACTS AND LOCATIONS:
Overall Officials: Shiow-Ching Shun, PhD, Principal Investigator — Department of Nursing, College of Medicine, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan